CLINICAL TRIAL: NCT03858972
Title: Multinational, Multicenter, Phase 2 Study of Tesetaxel Plus a Reduced Dose of Capecitabine in Patients With HER2 Negative, Hormone Receptor Positive, Locally Advanced or Metastatic Breast Cancer Who Have Not Previously Received a Taxane
Brief Title: Tesetaxel Plus Reduced Dose of Capecitabine in Patients With HER2 Negative, HR Positive, LA/MBC
Acronym: CONTESSA 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor has discontinued the development of tesetaxel
Sponsor: Odonate Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODO-TE-B201
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: Tesetaxel; Capecitabine; HER2 negative; Combination of tesetaxel and capecitabine; Taxane-naive; Locally advanced or metastatic breast cancer; Hormone receptor positive; Metastatic breast cancer (MBC); Breast cancer; Central nervous system (CNS) metastases; de novo metastatic breast cancer; Oral chemotherapy; Taxane
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — tesetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tesetaxel (oral) and capecitabine (oral) (Experimental): Cohort 1: Tesetaxel (27 mg/m2) once every 21 days on Day 1 of each 21-day cycle; and capecitabine (825 mg/m2) twice daily (total daily dose of 1,650 mg/m2) beginning with the evening dose on Day 1 through the morning dose on Day 15 of each 21-day cycle.
  Cohort 2: On Cycle 1, Day -1, either a single morning dose of capecitabine at 825 mg/m2 (Cohort 2A) or 1,250 mg/m2 (Cohort 2B). On Cycle 1, Day 1, a single dose of tesetaxel (27 mg/m2), followed 2 hours later by capecitabine (825 mg/m2), followed by an evening dose of capecitabine (825 mg/m2). Capecitabine (825 mg/m2) twice daily (total daily dose of 1,650 mg/m2) beginning with the morning dose on Day 2 through evening dose on Day 14 of Cycle 1. Starting with Cycle 2, tesetaxel (27 mg/m2) once every 21 days on Day 1 of each 21-day cycle; and capecitabine (825 mg/m2) twice daily (total daily dose of 1,650 mg/m2) beginning with the evening dose on Day 1 through the morning dose on Day 15 of each 21-day cycle.
  Interventions: Drug: Tesetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel plus reduced dose of capecitabine
Drug: Capecitabine — Reduced dose of capecitabine

SUMMARY:
CONTESSA 2 is a multinational, multicenter, Phase 2 study of tesetaxel in patients with HER2 negative, HR positive, locally advanced or metastatic breast cancer (LA/MBC) not previously treated with a taxane. The primary objective of the study is to establish the efficacy of tesetaxel plus a reduced dose of capecitabine based on objective response rate (ORR) as assessed by an Independent Radiologic Review Committee (IRC). 152 patients were enrolled.

DETAILED DESCRIPTION:
CONTESSA 2 is a multinational, multicenter, Phase 2 study of tesetaxel, an investigational, orally administered taxane, in patients with HER2 negative, HR Positive, LA/MBC not previously treated with a taxane in the neoadjuvant, adjuvant or metastatic setting. This Study complements CONTESSA, a multinational, multicenter, randomized, Phase 3 study in patients with HER2 negative, HR positive LA/MBC previously treated with a taxane in the neoadjuvant or adjuvant setting. 152 patients were enrolled, including 149 who received treatment. Patients are administered tesetaxel at 27 mg/m2 orally once every 21 days on the first day of each 21-day cycle plus capecitabine at 825 mg/m2 orally twice daily (for a total daily dose of 1,650 mg/m2) for 14 days of each 21-day cycle. Patients in the dense pharmacokinetics (PK) cohort receive a single dose of capecitabine monotherapy prior to starting the combination regimen. Capecitabine is an oral chemotherapy agent that is considered a standard-of-care treatment in LA/MBC. The primary efficacy endpoint is ORR as assessed by the IRC. The secondary efficacy endpoints are duration of response (DoR) as assessed by the IRC, progression-free survival (PFS) as assessed by the IRC, disease control rate (DCR) as assessed by the IRC and overall survival (OS). CONTESSA 2 also investigates the PK of tesetaxel.

ELIGIBILITY:
Inclusion criteria:

1. Female or male patients at least 18 years of age
2. Histologically or cytologically confirmed breast cancer
3. HER2 negative disease based on local testing: American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines should be utilized for assessing HER2 status
4. HR (ER and/or PgR) positive disease based on local testing: ASCO/CAP guidelines should be utilized for assessing HR status
5. Measurable disease per RECIST 1.1, including bone-only disease with measurable lytic component.

   Patients with bone-only metastatic cancer must have a measurable lytic or mixed lytic-blastic lesion that can be accurately assessed by computed tomography (CT) or magnetic resonance imaging (MRI). Patients with bone-only disease without a measurable lytic component (ie, blastic-only metastasis) are not eligible.

   Known metastases to the CNS are permitted but not required. The following criteria apply:
   * Patients must be neurologically stable and either off corticosteroids or currently treated with a maximum daily dose of 4 mg of dexamethasone (or equivalent), with no increase in corticosteroid dose within 7 days prior to Enrollment (defined as the time of Sponsor approval of treatment dose)
   * Patients with a history of CNS metastases but with no current evidence of CNS lesions following local therapy are eligible
   * Patients may have CNS metastases that are stable or progressing radiologically
   * Patients with current evidence of leptomeningeal disease are not eligible
   * Patients may have untreated brain metastases or previously treated brain metastases, as long as no immediate local CNS-directed therapy is indicated
   * Any prior whole brain radiation therapy must have been completed > 14 days prior to the date of Enrollment
   * Prior stereotactic brain radiosurgery is permitted
   * CNS surgical resection must have been completed > 28 days prior to the date of Enrollment; patient must have complete recovery from surgery
6. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
7. Prior endocrine therapy with or without a CDK 4/6 inhibitor unless endocrine therapy is not indicated (ie, short relapse-free interval while on adjuvant endocrine therapy [endocrine resistance]; rapidly progressing disease/visceral crisis; or endocrine intolerance). Any targeted therapies approved for HER2 negative, HR positive LA/MBC, including everolimus, are permitted as prior therapy. There is no limit to the number of prior endocrine therapies.
8. Documented (including de novo): (a) locally advanced breast cancer that is not considered curable by surgery and/or radiation; or (b) metastatic breast cancer
9. Adequate hematologic, hepatic and renal function, as evidenced by:

   * Absolute neutrophil count (ANC) ≥ 1,500/μL without colony-stimulating factor support
   * Platelet count ≥ 100,000/μL
   * Hemoglobin ≥ 10 g/dL without need for hematopoietic growth factor or transfusion support
   * Total bilirubin < 1.5 × upper limit of normal (ULN); does not apply to patients with Gilbert's syndrome
   * Alanine aminotransferase (ALT) < 3 × ULN unless hepatic metastases are present then < 5 × ULN
   * Aspartate aminotransferase (AST) < 3 × ULN unless hepatic metastases are present then < 5 × ULN
   * Alkaline phosphatase < 2.5 × ULN unless hepatic metastases are present then < 5 × ULN
   * Calculated creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula or local standard)
   * Serum albumin ≥ 3.0 g/dL
   * Prothrombin time (PT) < 1.5 × ULN or international normalized ratio (INR) < 1.3 and partial thromboplastin time (PTT) < 1.5 × ULN, unless the patient is on a therapeutic anticoagulant
10. Complete recovery to baseline or Grade 1 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 from adverse effects of prior surgery, radiotherapy, endocrine therapy, and other therapy, as applicable, with the exception of Grade 2 alopecia from prior chemotherapy
11. Ability to swallow an oral solid-dosage form of medication
12. A negative serum pregnancy test within 7 days prior to the first dose of Study treatment in women of childbearing potential (ie, all women except those who are post menopause for ≥ 1 year or who have a history of hysterectomy or surgical sterilization)
13. Women of childbearing potential must use an effective, non-hormonal form of contraception from Screening throughout the Treatment Phase and until 70 days after the last dose of Study treatment

    * Acceptable methods include: copper intrauterine device or double barrier methods, including male/female condoms with spermicide and use of contraceptive sponge, cervical cap, or diaphragm
14. Male patients must use an effective, non-hormonal form of contraception from Screening throughout the Treatment Phase and until 130 days after the last dose of Study treatment

    * Acceptable methods include: male/female condoms with spermicide, or vasectomy with medical confirmation of surgical success
15. Written informed consent and authorization to use and disclose health information
16. Ability to comprehend and comply with the requirements of the Study

Exclusion criteria:

1. Two or more prior chemotherapy regimens for advanced disease
2. Prior treatment with a taxane at any dose
3. Prior treatment with capecitabine at any dose
4. Current evidence of leptomeningeal disease
5. Other cancer that required therapy within the preceding 5 years other than adequately treated: (a) non-melanoma skin cancer or in situ cancer; or (b) following approval by the Medical Monitor, other cancer that has a very low risk of interfering with the safety or efficacy endpoints of the Study
6. Known human immunodeficiency virus infection, unless well controlled. Patients who are on an adequate antiviral regimen with no evidence of active infection are considered well controlled.
7. Active hepatitis B or active hepatitis C infection
8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with Study participation or investigational product administration or may interfere with the interpretation of Study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this Study.
9. Presence of neuropathy > Grade 1 per NCI CTCAE version 5.0
10. Anticancer treatment, including endocrine therapy, radiotherapy (except stereotactic brain radiosurgery), chemotherapy, biologic therapy, or therapy in an investigational clinical study, ≤ 14 days prior to the date of Enrollment
11. Major surgery ≤ 28 days prior to the date of Enrollment; patient must have complete recovery from surgery
12. Less than 2 weeks or 5 plasma half-lives (whichever is greater) since last use of a medication or ingestion of an agent, beverage, or food that is a known clinically relevant strong inhibitor or known clinically relevant inducer of the cytochrome P450 (CYP)3A pathway (patients should discontinue taking any regularly-taken medication that is a strong inhibitor or inducer of the CYP3A pathway)
13. History of hypersensitivity or unexpected reactions to capecitabine, fluoropyrimidine agents or any of their ingredients
14. Known dihydropyrimidine dehydrogenase (DPD) deficiency. Testing for DPD deficiency must be performed where required by local regulations, using a validated method that is approved by local health authorities.
15. Pregnant or breastfeeding
16. If, in the opinion of the Investigator, the patient is deemed unwilling or unable to comply with the requirements of the Study
17. Treatment with brivudine, sorivudine, or its chemically-related analogs ≤ 28 days prior to the date of Enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
ORR as assessed by the IRC | Approximately 2.0-2.5 years

SECONDARY OUTCOMES:
DoR as assessed by the IRC | Approximately 2.0-2.5 years
PFS as assessed by the IRC | Approximately 2.0-2.5 years
DCR as assessed by the IRC | Approximately 2.0-2.5 years
OS | Approximately 3.0-3.5 years
Central nervous system (CNS) ORR as assessed by the CNS IRC in patients with CNS metastases at baseline | Approximately 2.0-2.5 years
CNS DoR as assessed by the CNS IRC in patients with CNS metastases at baseline | Approximately 2.0-2.5 years
CNS PFS as assessed by the CNS IRC in patients with CNS metastases at baseline or a history of CNS metastases and in the intent-to-treat (ITT) population | Approximately 2.0-2.5 years
CNS OS in patients with CNS metastases at baseline or a history of CNS metastases | Approximately 3.0-3.5 years

OTHER OUTCOMES:
Adverse events, including deaths and other serious adverse events | Approximately 3.0-3.5 years
Incidence of clinical laboratory abnormalities (e.g., CBC, serum chemistry and coagulation testing) | Approximately 3.0-3.5 years
Peak plasma concentration (Cmax) of tesetaxel | Approximately 2.0-2.5 years
Area under the plasma concentration versus time curve (AUC) of tesetaxel | Approximately 2.0-2.5 years
The effect of tesetaxel on capecitabine and 5-FU Cmax | Approximately 2.0-2.5 years
The effect of tesetaxel on capecitabine and 5-FU AUC | Approximately 2.0-2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Connell, MD, Study Director — Odonate Therapeutics, Inc.
Locations (25):
- United States (9):
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Center, Lakewood, Colorado
  - Sarah Cannon Research Institute - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New York Cancer and Blood Specialists, East Setauket, New York
  - West Cancer Center, Germantown, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Border Medical Oncology, Albury, New South Wales, Australia
- Canada (6):
  - Hopital Maisonneuve-Rosemont, Montreal
  - Center Hospitalier de Montreal CHUM McPeak Sirois, Montreal
  - CIUSSS de Centre-Ouest-de-l'Île-de-Montréal Jewish General Hospital, Montreal
  - McGill University Health Center, Montreal
  - CHU de Quebec-University Laval, Québec
  - Centre Hospitalier Universitaire de Sherbrooke CIUSSS de lEstrie CHUS patyre, Sherbrooke
- South Korea (5):
  - Kyungpook National University Hospital, Daegu
  - National Cancer Center, Goyang
  - Gangnam Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (2):
  - Hospital Teresa Herrera Materno-Infantil (CHUAC), A Coruña
  - Fundacion Jimenez Diaz, Madrid
- Taiwan (2):
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei